CLINICAL TRIAL: NCT05262270
Title: Randomized, Placebo-Controlled Trial of Extended-Release Naltrexone and Monthly Extended-Release Buprenorphine for Cocaine Use Disorder (CURB-2)
Brief Title: Extended-Release Naltrexone and Monthly Extended-Release Buprenorphine for Cocaine Use Disorder (CURB-2)
Acronym: CURB-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, MD, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU-2021-0223; UG1DA020024 (NIH)
Record Dates: First submitted 2022-02-17; First posted 2022-03-02 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Cocaine Use Disorder
Keywords: Naltrexone; Buprenorphine; Extended release injectable Naltrexone; Extended release injectable Buprenorphine; CUD; Cocaine; Cocaine Abuse
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — phospholamban

STUDY DESIGN:
Intervention Model Description: The study intervention is three doses of 380mg XR-NTX (Weeks 0, 3 and 6) and two doses of 300mg XR-BUP (Weeks 0, 4). XR-NTX is delivered via intramuscular (IM) injection in the gluteus; XR-BUP is delivered via subcutaneous (SQ) injection in the abdomen.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind, placebo-controlled study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug intervention (XR-NTX+XR-BUP) (Experimental): The study intervention is three doses of 380mg XR-NTX (Weeks 0, 3 and 6) and two doses of 300mg XR-BUP (Weeks 0, 4).
  Drug: XR-NTX XR-NTX: 3 intramuscular injections administered Week 0, 3, 6. Other Names: Extended Release Injectable Naltrexone Arm: Experimental
  Drug: XR-BUP XR-BUP: 2 subcutaneous injections administered Week 0, 4. Other Names: Extended Release Injectable Buprenorphine Arm: Experimental
  Interventions: Drug: Extended-Release Naltrexone; Drug: Extended Release Buprenorphine
- Placebo (Placebo Comparator): Matched placebo injections (PBO-Inj) for the treatment of cocaine use disorder (CUD).
  Drug: Placebo (PLB) Injectable Placebo: 3 intramuscular injections administered Week 0, 3, 6. Other Names: Injectable matching (to XR-NTX) placebo Arm: Placebo Comparator - matched Placebo (PLB)
  Drug: Placebo (PLB) Injectable Placebo: 2 subcutaneous injections administered Week 0, 4. Other Names: Injectable matching (to XR-BUP) placebo Arm: Placebo Comparator - matched Placebo (PLB)
  Interventions: Drug: Placebo (PLB) Injectable matched to XR-NTX; Drug: Placebo (PLB) Injectable matched to XR-BUP

INTERVENTIONS:
Drug: Extended-Release Naltrexone — XR-NTX (Extended-Release Naltrexone) doses of 380mg (Weeks 0, 3 and 6) via intramuscular (IM) injections in the gluteus.
  Other Names: XR-NTX
  Arms: Drug intervention (XR-NTX+XR-BUP)
Drug: Extended Release Buprenorphine — Extended-Release buprenorphine (XR-BUP) two doses of 300mg XR-BUP (Weeks 0, 4) via subcutaneous injections in the abdomen. Option for 100mg at Weeks 3 and 6 (if needed to alleviate side effects).
  Other Names: XR-BUP
  Arms: Drug intervention (XR-NTX+XR-BUP)
Drug: Placebo (PLB) Injectable matched to XR-NTX — 3 doses of intramuscular injections (Week 0, 3, 6)
  Other Names: Injectable matching (to XR-NTX) placebo
  Arms: Placebo
Drug: Placebo (PLB) Injectable matched to XR-BUP — 2 doses of subcutaneous injections (Week 0, 4)
  Other Names: Injectable matching (to XR-BUP) placebo
  Arms: Placebo

SUMMARY:
This is an 8-week, double-blind, randomized placebo-controlled trial of the efficacy of a combination of extended-release naltrexone (XR-NTX) and extended-release buprenorphine (XR-BUP) compared to matched placebo injections (PBO-Inj) for the treatment of cocaine use disorder (CUD).

DETAILED DESCRIPTION:
The primary objective of this study is to assess the efficacy of XR-NTX plus XR-BUP as a combination pharmacotherapy for CUD. Approximately four hundred and twenty-six adults will be randomized into the study at 8-12 sites in the U.S. Eligibility will be determined during a maximum 21-day screening period. After screening/baseline is completed and eligibility is confirmed, participants will be randomized and begin the 1-week medication induction phase followed by the 8-week medication phase of the trial.

Participants will be randomized in a 1:1 ratio to either 1) XR-NTX + XR-BUP arm and receive injections of extended-release naltrexone (XR-NTX; as Vivitrol®) and extended-release buprenorphine (XR-BUP; as SublocadeTM), or to 2) PBO-Inj matching the timeline and delivery methods of injections for the XR-NTX + XR-BUP arm. XR-NTX or PBO-Inj injections will be provided on the day of randomization and in Weeks 3 and 6. XR-BUP or PBO-Inj injections will be provided on days 3-5 following randomization and in week 4. During the 1-week induction phase and the 8-week medication phase, participants will be asked to attend clinic twice weekly for collection of urine samples and to complete assessments as indicated on the schedule of assessments. Following the 8-week medication phase, participants will be asked to attend clinic weekly for the follow-up phase during Weeks 9-12.

Participants will be involved in the study for approximately 16 weeks, including a screening/baseline period of up to 3 weeks (i.e., 21 days), 1 week for randomization and medication induction, 8 weeks of medication, and 4 weeks of follow-up. The screening phase may differ by participant in the length of time needed to complete preliminary eligibility assessments. Randomization and medication induction visit may take approximately 2 hours. Twice-weekly visits during the medication phase will range from about 20 to 90 minutes in length depending on scheduled assessments. Medication administration visits may require an additional 2 hours. Visits in the follow-up phase will take place approximately 30-60 minutes to complete. An 8-week medication period was selected based on expected time for group differences to emerge and for pragmatic issues related to medication dosing.

Enrollment is expected to take place over a period of approximately 13 months, with an approximate total of 16 months of study visits.

ELIGIBILITY:
Individuals must meet all of the inclusion criteria and no exclusion criteria in order to be eligible to participate in the study, including but not limited to:

Inclusion Criteria:

1. Be 18 to 65 years of age;
2. Be interested in reducing or stopping cocaine use.
3. Be willing to comply with all study procedures and medication instructions.

Exclusion Criteria:

1. Have any condition for which, in the opinion of the site investigator or designee, study participation would not be in their best interest or that could prevent, limit, or confound the protocol-specified assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
Proportion of Cocaine-negative UDS | Week 5 up to Week 8
  The primary outcome measure is the proportion of cocaine-negative UDS obtained during Weeks 5 through 8 of the medication phase as measured for the XR-NTX + XR-BUP and PBO-Inj conditions. The primary outcome (UDS) has been chosen because it is an objective measure of cocaine use and was the outcome showing significant improvement over placebo in the original CURB trial.

SECONDARY OUTCOMES:
Number of participants who Self-report cocaine use | 8 Weeks
  Self-report elicited through Timeline Followback (TLFB) on days of cocaine use during Weeks 0-8;
Mean self reported cocaine craving score | 8 Weeks
  Cocaine craving as measured by the Visual Analog Craving Scales (VAS) during Weeks 0-8.
  Possible scores range from 0 to 100, with higher scores indicating worse craving.
Measures of safety (adverse events) | 8 weeks
  Number and severity of adverse events reported during Weeks 0-8; Number and outcomes (non-fatal and fatal) of overdose events during Weeks 0-8
Mean self reported overall functioning | Week 8
  Self-report overall functioning as measured by the Treatment Effectiveness Assessment (TEA) at Week 8. Possible scores range from 1 to 10 for each of the 4 domains, with higher scores indicating better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar Trivedi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (12):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UCLA Vine Street Clinic, Los Angeles, California
  - Center on Substance Use and Health (CSUH), San Francisco, California
  - Cove Behavioral Health, Tampa, Florida
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Mountain Manor Treatment Center, Baltimore, Maryland
  - Berman Center for Outcomes and Clinical Research at Hennepin Healthcare, Minneapolis, Minnesota
  - Addictions Institute of Mount Sinai, New York, New York
  - UTSW Medical Center, Center for Depression Research and Clinical Care, Dallas, Texas
  - University of Texas Health San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be available to researchers on the website https://datashare.nida.nih.gov/ after the study is complete and the data is analyzed. This website will not include information that can identify individual study participants. The following information will be posted: Study protocol, reference to study publication of primary outcome, data sets (SAS and ASCII ), annotated case report forms, define file (also known as Data Dictionary), study-specific de-identification notes. Prior to downloading any study data, the user will be prompted to complete a registration agreement for data use. Users will have to register a name and valid e-mail address in order to download data and to accept their responsibility for using data in accordance with the National Institute on Drug Abuse (NIDA) Data Share Agreement.
Supporting Information: Study Protocol, CSR
Time Frame: This will be available five months after all sites are closed. No yet determined duration of availability.
Access Criteria: Researchers who are active users on the https://datashare.nida.nih.gov/ site. Primary data will be available to the public in the NIDA data repository on this site as well.
URL: https://datashare.nida.nih.gov/

REFERENCES:
- [Background] Center for Behavioral Health Statistics and Quality. 2019 National Survey on Drug Use and Health (NSDUH): CAI Specifications for Programming (English Version). Substance Abuse and Mental Health Services Administration, editor. Rockville, MD; 2018.
- [Background] Czoty PW, Stoops WW, Rush CR. Evaluation of the "Pipeline" for Development of Medications for Cocaine Use Disorder: A Review of Translational Preclinical, Human Laboratory, and Clinical Trial Research. Pharmacol Rev. 2016 Jul;68(3):533-62. doi: 10.1124/pr.115.011668. PMID 27255266
- [Background] Whitfield TW Jr, Schlosburg JE, Wee S, Gould A, George O, Grant Y, Zamora-Martinez ER, Edwards S, Crawford E, Vendruscolo LF, Koob GF. kappa Opioid receptors in the nucleus accumbens shell mediate escalation of methamphetamine intake. J Neurosci. 2015 Mar 11;35(10):4296-305. doi: 10.1523/JNEUROSCI.1978-13.2015. PMID 25762676
- [Background] Ling W, Hillhouse MP, Saxon AJ, Mooney LJ, Thomas CM, Ang A, Matthews AG, Hasson A, Annon J, Sparenborg S, Liu DS, McCormack J, Church S, Swafford W, Drexler K, Schuman C, Ross S, Wiest K, Korthuis PT, Lawson W, Brigham GS, Knox PC, Dawes M, Rotrosen J. Buprenorphine + naloxone plus naltrexone for the treatment of cocaine dependence: the Cocaine Use Reduction with Buprenorphine (CURB) study. Addiction. 2016 Aug;111(8):1416-27. doi: 10.1111/add.13375. Epub 2016 Apr 21. PMID 26948856
- [Background] Trivedi MH, Wisniewski SR, Morris DW, Fava M, Kurian BT, Gollan JK, Nierenberg AA, Warden D, Gaynes BN, Luther JF, Rush AJ. Concise Associated Symptoms Tracking scale: a brief self-report and clinician rating of symptoms associated with suicidality. J Clin Psychiatry. 2011 Jun;72(6):765-74. doi: 10.4088/JCP.11m06840. PMID 21733477
- [Background] dela Cruz AM, Bernstein IH, Greer TL, Walker R, Rethorst CD, Grannemann B, Carmody T, Trivedi MH. Self-rated measure of pain frequency, intensity, and burden: psychometric properties of a new instrument for the assessment of pain. J Psychiatr Res. 2014 Dec;59:155-60. doi: 10.1016/j.jpsychires.2014.08.003. Epub 2014 Aug 27. PMID 25194231
- [Background] Ling W, Farabee D, Liepa D, Wu LT. The Treatment Effectiveness Assessment (TEA): an efficient, patient-centered instrument for evaluating progress in recovery from addiction. Subst Abuse Rehabil. 2012 Jan 1;3(1):129-136. doi: 10.2147/SAR.S38902. PMID 23580868
- [Background] Pettinati HM, Kampman KM, Lynch KG, Suh JJ, Dackis CA, Oslin DW, O'Brien CP. Gender differences with high-dose naltrexone in patients with co-occurring cocaine and alcohol dependence. J Subst Abuse Treat. 2008 Jun;34(4):378-90. doi: 10.1016/j.jsat.2007.05.011. Epub 2007 Jul 30. PMID 17664051
- [Background] Nasser AF, Heidbreder C, Liu Y, Fudala PJ. Pharmacokinetics of Sublingual Buprenorphine and Naloxone in Subjects with Mild to Severe Hepatic Impairment (Child-Pugh Classes A, B, and C), in Hepatitis C Virus-Seropositive Subjects, and in Healthy Volunteers. Clin Pharmacokinet. 2015 Aug;54(8):837-49. doi: 10.1007/s40262-015-0238-6. PMID 25603822
- [Background] Winhusen TM, Kropp F, Lindblad R, Douaihy A, Haynes L, Hodgkins C, Chartier K, Kampman KM, Sharma G, Lewis DF, VanVeldhuisen P, Theobald J, May J, Brigham GS. Multisite, randomized, double-blind, placebo-controlled pilot clinical trial to evaluate the efficacy of buspirone as a relapse-prevention treatment for cocaine dependence. J Clin Psychiatry. 2014 Jul;75(7):757-64. doi: 10.4088/JCP.13m08862. PMID 24911028
- [Background] Kariisa M, Scholl L, Wilson N, Seth P, Hoots B. Drug Overdose Deaths Involving Cocaine and Psychostimulants with Abuse Potential - United States, 2003-2017. MMWR Morb Mortal Wkly Rep. 2019 May 3;68(17):388-395. doi: 10.15585/mmwr.mm6817a3. PMID 31048676
- [Derived] Trivedi MH, Kalmin MM, Carmody T, Chongsi EM, Ghitza UE, Jha MK, Mayes TL, Casey-Willingham A, Sethuram S, Marino EN, Monastirsky M, Shoptaw SJ. Randomized, placebo-controlled trial of injectable extended-release naltrexone and injectable extended-release buprenorphine for cocaine use disorder (CURB-2): Study rationale and design. Contemp Clin Trials. 2025 Jul;154:107954. doi: 10.1016/j.cct.2025.107954. Epub 2025 May 11. PMID 40360074

DOCUMENTS (5):
  • Informed Consent Form: Part 1 - For All sites and California site (2024-10-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT05262270/ICF_000.pdf
  • Informed Consent Form: Part-2- For UCSF site (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/70/NCT05262270/ICF_001.pdf
  • Informed Consent Form: Part 2- For UIC site (2024-11-11): https://cdn.clinicaltrials.gov/large-docs/70/NCT05262270/ICF_002.pdf
  • Informed Consent Form: Part 2- For Mt. Sinai site (2024-11-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT05262270/ICF_003.pdf
  • Informed Consent Form: Part 2- For Rest of the sites including UTSW (lead site) (2024-05-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT05262270/ICF_004.pdf